CLINICAL TRIAL: NCT05169957
Title: Hepatic Ablation of Melanoma Metastases to Enhance Immunotherapy Response, a Phase I Clinical Trial (HAMMER I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2021.036; HUM00201698 (Other: University of Michigan)
Record Dates: First submitted 2021-12-09; First posted 2021-12-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Melanoma, Ocular; Melanoma, Cutaneous; Metastatic Melanoma; Melanoma, Mucosal; Liver Metastases
Keywords: Liver SBRT; ipilimumab; nivolumab
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Ipilimumab; Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab + Nivolumab + Stereotactic Body Radiation Therapy (SBRT) (Experimental): Liver SBRT following the second cycle of ipilimumab + nivolumab, which will then be continued up to 4 total cycles prior to subsequent maintenance nivolumab for duration of clinical benefit and tolerance (standard of care systemic therapy)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Procedure: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab administered IV over 85-100 minutes at 3 mg/kg (combined with nivolumab administered IV over 30-60 minutes at 1 mg/kg) every 3 weeks for a total of 4 doses or until progression or unacceptable toxicity.
Drug: Nivolumab — Nivolumab administered IV over 30-60 minutes at 1 mg/kg (combined with ipilimumab administered IV over 85-100 minutes at 3 mg/kg) every 3 weeks for a total of 4 doses of the combination therapy or until progression or unacceptable toxicity. Subjects may receive maintenance dosing of nivolumab alone administered IV over 30-60 minutes at 240 mg every 2 weeks or 480 mg every 4 weeks for a maximum of 52 weeks or until progression or unacceptable toxicity.
Procedure: Stereotactic Body Radiation Therapy — 24-45 Gy delivered in three fractions to up to 4 liver metastases
  Other Names: SBRT

SUMMARY:
The primary purpose of this study is to determine the feasibility of liver stereotactic body radiation therapy (SBRT) given in combination with systemic therapy (ipilimumab and nivolumab) in adults with metastatic melanoma with liver metastases who are at significant risk of not benefiting from systemic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) with histologically or cytologically confirmed metastatic melanoma for which surgery is not recommended with liver metastases; disease must be measurable per RECIST criteria
* Patients must have a life expectancy of at least 6 months
* Patients must have a performance status of 0 - 2 on the ECOG Performance Scale.
* Allowable prior therapy:

  * Previous adjuvant or neoadjuvant treatment for melanoma is allowed, which may include molecularly-targeted agents, IFN-alpha, ipilimumab, nivolumab, and pembrolizumab, if it was completed at least 6 weeks before enrollment in the study.
  * Patients who had experienced treatment-related adverse events from prior adjuvant or neoadjuvant treatment for melanoma are allowed if symptoms had returned to baseline or had stabilized.
  * Prior stereotactic radiotherapy (SBRT) of extrahepatic metastases is permitted.
* Patients must be willing to undergo multiple liver tissue biopsies
* Patients must have adequate organ function per protocol
* Patients must understand and be willing to sign an informed consent form approved for this purpose by the Institutional Review Board (IRB) of the University of Michigan Medical Center indicating that they are aware of the investigational aspects of the treatment and the potential risks.
* Participants of childbearing potential

  * Female subject of childbearing potential should have a serum pregnancy within 14 days of enrollment and 72 hours prior to receiving the first dose of I/N, and must be willing to use a highly effective method of contraception for the course of the study through 180 days after the last dose of I/N. (Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.)
  * Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 180 days after the last dose of study therapy. Sperm donation is prohibited while on study. (Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.)

Exclusion Criteria:

* Patients will be excluded from the trial if participants have the following:
* Diffuse involvement of liver by cancer on CT, PET, or MRI imaging
* More than 4 liver metastases on CT scan at time of initial assessment. If a flare occurs during the initial I/N cycles, up to 8 metastases may be targeted if able to be targeted by a minimum of 8 Gy per fraction while meeting normal tissue constraints.
* Diagnosis of underlying parenchymal end stage liver disease (cirrhosis) or biliary disease (primary biliary cirrhosis).
* Other locally advanced or metastatic invasive malignancy active within last 3 years, excluding in situ or localized cancers or malignancies which have been treated
* Patients who had received previous systemic anticancer therapy for unresectable or metastatic melanoma
* Has known active carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least two weeks prior to enrollment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to enrollment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

  • Note: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Require daily corticosteroids >10 mg of prednisone (or its equivalent)

  * Note: Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would NOT be excluded from the study.
  * Note: Patients who require the use of topical steroids would not be excluded.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with informed consent through 180 days after the last dose of trial treatment.
* Has a diagnosis of immunodeficiency (including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency (AIDS)-related illness) or has received a bone marrow transplant or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has known active Hepatitis B or Hepatitis C.
* Prior Gr3/4 life threatening immune related adverse event that is considered an unacceptable risk per the treating investigator
* Has received a live vaccine within 30 days of enrollment.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
  * COVID vaccination acceptable; preferably all doses administered 7 days prior to start of therapy
* Lacks insurance preapproval for SBRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who receive all planned radiotherapy. | Up to 5 weeks after start of study treatment
  Percentage of patients who receive all fractions of radiotherapy as planned following the second cycle of ipilimumab/nivolumab (I/N). Radiotherapy will be administered on C2D8 of I/N (±7days)

SECONDARY OUTCOMES:
Proportion of patients who develop grade 3 or higher toxicity | Up to 14 weeks after start of study treatment
  Proportion of patients who develop grade three or higher toxicities within 60 days after treatment with SBRT or thirty days after the last cycle of I/N, whichever occurs later. Any serious adverse event that occurs after this time frame and is considered related to the study treatment will also be reported.
Overall survival (OS) | Up to 2 years after end of study treatment
  OS defined as the time from start of treatment to death. This will be analyzed using Kaplan-Meier curves and descriptive statistics.
Progression free-survival (PFS) | Up to 2 years after end of study treatment
  PFS defined as the time from start of treatment to date of radiological or clinical progression (leading to withdrawal from the study), or death from any cause, whichever comes first. Assessed Per RECIST v1.1; analyzed using Kaplan-Meier curves and descriptive statistics.
Proportion of patients with local control | Up to 2 years after end of study treatment
  Freedom from local progression (local control) is defined as the lack of progression of the tumors treated by RT, either by tumor size or enhancement. Progression or development of new tumors elsewhere in the liver or outside of the liver would not constitute a local control failure. Tumors which increase in size or demonstrate new or increasing enhancement are considered progression. Analyzed using Kaplan-Meier curves and descriptive statistics.
Objective response rate (ORR) | Up to 2 years after end of study treatment
  The percentage of patients whose disease decreases (Partial response - PR) and/or disappears (Complete response - CR) after treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Best overall response (BoR) | Up to 2 years after end of study treatment
  The best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Green, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No